CLINICAL TRIAL: NCT00694668
Title: The (Cost-) Effectiveness of Mindfulness-training and Cognitive Behavioural Therapy in Adolescents and Young Adults With Deliberate Self Harm
Acronym: DSH
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); University Medical Centre Nijmegen(departement of psychiatry) (Unknown)
Responsible Party: Anne van Giezen, PhD, Leiden University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 120610008
Record Dates: First submitted 2008-06-05; First posted 2008-06-10 (Estimated); Last update posted 2009-11-06 (Estimated); Status verified 2009-11

CONDITIONS: Self-Injurious Behavior
Keywords: Deliberate Self-Harm; Self-Injurious Behaviour; Suicidal Behaviour; Cognitive behavioural therapy; Mindfulness Based cognitive therapy
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Cognitive Behavioural Treatment
  Interventions: Behavioral: Cognitive Behavioral treatment
- 2 (Experimental): Mindfulness Based Cognitive Therapy-training
  Interventions: Behavioral: Mindfulness based cognitive therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral treatment — Brief cognitive behavioral therapy (12 sessions)
  Arms: 1
Behavioral: Mindfulness based cognitive therapy — 9 sessions MBCT in a group-format (up to 8 persons)
  Arms: 2

SUMMARY:
Background:

In recent years, there has been a marked rise in the frequency of young people engaging in Deliberate Self-Harm (DSH). DSH refers to all kinds of self-harming behaviour, with and without suicidal intent. Early identification and treatment of persons who engaged in DSH is important because every episode of DSH increases the risk of future episodes and, eventually, suicide. A number of comprehensive treatment programs have been developed and proven to be effective in reducing DSH in adults. Especially the modification of inadequate emotion regulation strategies seems to be essential in the prevention of future episodes of DSH. The first short-term results of a Dutch time-limited and structured individual cognitive-behavioral treatment (CBT) for DSH in adolescents and young adults also showed positive effects on repetition of DSH and associated problems.

Objective:

To study the effects and costs of the total individual CBT package and one of the components of the total CBT treatment package (i.e. mindfulness training) in a group format compared to Treatment-as-Usual (TAU) on the short and long term.

Design:

Multi-center randomized controlled clinical trial with repeated measurements at baseline (M0),and posttreatment (M6)), 12 (M12) and 18 months (M18) after baseline.

Procedure:

Young persons aged 15-35 who recently have engaged in DSH and have been referred to the Leiden University Medical Centre, the mental health centre Rivierduinen or the University Medical Centre St. Radboud following an act of DSH will be invited to participate. Persons reporting severe psychiatric disorders requiring intensive inpatient treatment or serious cognitive impairments will be excluded.

Interventions:

Participants are randomly allocated to CBT, Mindfulness-Based Cognitive Therapy(MBCT) or Treatment-as-Usual (TAU). The CBT treatment consists of up to 12 weekly sessions of individual treatment mainly consisting of emotion regulations skills, cognitive restructuring, and behavioural skills training. The MBCT training consists of 8 2-hour sessions in a group format within a three months time frame.

Outcome measures:

The same outcome measures to assess the clinical effects of treatment as in the previous study will be used (repetition of DSH, depression (BDI-II), anxiety (SCL-90), self-concept(RSC-Q), and suicide cognitions (SCS)) allowing a historical comparison of treatment effectiveness across both randomized clinical trials. In addition at all assessments health-related quality of life, use of medical resources and loss of productivity will be assessed (EuroQol, VAS and TTO). In addition,problems in emotion regulation (an important risk mechanism for repetition of DSH) will be assessed before and after treatment.

Economic evaluation:

Differences in societal costs (intervention, other (health) care and productivity)will be compared to differences in the frequency of DSH and quality adjusted life years (EuroQol, VAS and TTO).

Data-analysis/power:

Based on our previous study at least a medium effect of treatment on repetition of DSH may be expected. Assuming a medium effect of one of the treatments compared to TAU (delta =.75) and an attrition rate of about 20 %, at least 42 patients per study arm are needed to detect a minimal clinical relevant difference in repetition of DSH with a power of 80% and alpha set at .05.

ELIGIBILITY:
Inclusion Criteria:

* Recently engaged in an act of DSH including overdose of medication, ingestion of chemical substances and self-inflicted injuries according to the definition which is used in the WHO/Euro Multicentre Study on parasuicide:"An act with non-fatal outcome in which an individual deliberately initiates a non-habitual behavior, that without intervention from other will cause self-harm, or deliberately ingests a substance in excess of the prescribed or generally recognized dosage, and which is aimed at realizing changes that the person desires via the actual or expected physical consequences"(Platt et al., 1992).
* Aged between 15 and 35
* Living in the region of Leiden or Nijmegen

Exclusion Criteria:

* Severe psychiatric disorder or substance abuse requiring intensive inpatient treatment
* Serious cognitive impairments
* Not be able to converse in Dutch

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-11 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Repetition of DSH, measured by the suicide attempt and self injury interview (SASII). Frequency, method and other characteristics of deliberate self-harm and suicide attempts are assessed. | M0, M6, M12, M18

SECONDARY OUTCOMES:
depression, as measured by the Beck depression Inventory II | M0, M6, M12, M18
Anxiety, as measured by the symptom checklist '90 | M0, M6, M12, M18
Hostility, as measured by the symptom checklist '90 | M0, M6, M12, M18
Self-concept, as measured by the Robson self-concept questionnaire | M0, M6, M12, M18
Suicidal cognitions, as measured by the suicidal cognitions scale | M0, M6, M12, M18
QALYs, assessed by the EQ5D | M0, M6, M12, M18
COSTS, assessed by a 6-monthly diary | M0 - M6, M6 - M12, M12 - M18
Problem-solving skills, as measured by the Means Ends Problem-Solving Test | M0, M6
Experimental avoidance, as measured by the Acceptance and Action Questionnaire | M0, M6
difficulties in emotion-regulation, as measured by the difficulties in emotion regulation scale | M0, M6
general tendency to ruminate, as measured by the Ruminative Response Scale | M0, M6
mindfulness skills, as measured by the Five Facet Mindfulness Questionnaire | M0, M6
pathological dissociation, as measured by the dissociative experiences scale - taxon | M0, M6
Autobiographical memory, assessed by the autobiographical memory task | M0, M6
worrying, as measured by the Penn State Worry Questionnaire | M0 M6

CONTACTS AND LOCATIONS:
Overall Officials: Philip Spinhoven, Prof. dr., Study Chair — Leiden University, Institute for Psychological Research; Arnold A.P. van Emmerik, Dr., Study Director — Leiden University, Clinical Psychology Unit; Anne E. van Giezen, Dr., Study Director — Leiden University, Institute for Psychological Research, Clinical Psychology Unit; Anne E.M. Speckens, Prof. dr., Study Chair — Radboud University Medical Center; Suzanne de Klerk, MSc., Principal Investigator — Leiden University, Institute for Psychological Research, Clinical Psychology Unit
Locations (3):
- Netherlands (3):
  - University Medical Centre St. Radboud, Nijmegen, Gelderland
  - Leiden University Medical Centre, Leiden, South Holland
  - Rivierduinen Mental Health Centre, Leiden, South Holland